CLINICAL TRIAL: NCT00193076
Title: A Phase II Trial of Combination Gemcitabine, Carboplatin With or Without Trastuzumab in Patients With Metastatic Breast Cancer
Brief Title: Combination Gemcitabine, Carboplatin With or Without Trastuzumab in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Eli Lilly and Company (Industry); Genentech, Inc. (Industry)
Responsible Party: Denise A. Yardley, M.D., Sarah Cannon Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 63; B9E-US-S324; H3036S; NCT00191776 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Carboplatin; Trastuzumab

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine
Drug: Carboplatin — Carboplatin
Drug: Trastuzumab — Trastuzumab

SUMMARY:
Pre-clinical data suggests that combination therapy with gemcitabine and carboplatin is synergistic, and both drugs may be synergistic with trastuzumab. Additionally, recent clinical data suggest that the combination of gemcitabine with platinum is an active regimen in metastatic breast cancer. This study will test the combination of gemcitabine with carboplatin in patients with metastatic breast cancer. Patients with Her2/neu overexpression will be stratified to receive trastuzumab in addition to gemcitabine and carboplatin.

DETAILED DESCRIPTION:
Upon determination of eligibility, all patients will receive the following treatment:

Gemcitabine + Carboplatin

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Locally advanced or metastatic breast cancer
* Measurable disease as per RECIST criteria
* No prior chemotherapy in the metastatic breast setting
* Prior chemotherapy and/or hormonal therapy for early stage breast cancer
* Adjuvant Herceptin is allowed
* Prior radiation therapy in either the metastatic or early stage setting
* Patients may have received any number of hormonal therapies
* Age >18 years
* Only women are eligible for the study
* Able to perform activities of daily living with minimal assistance
* Normal organ and bone marrow function
* Patients who will be receiving Trastuzumab must have normal heart function
* Sign a written informed consent document

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Received prior chemotherapy for metastatic breast cancer
* Known leptomeningeal carcinomatosis
* Uncontrolled brain metastasis
* Uncontrolled intercurrent illness
* Pregnant or lactating
* History of other non-breast cancer malignancy
* Received prior chemotherapy for early stage breast cancer within 6 months

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2003-11; Primary Completion 2006-05 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Overall response rates | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Denise A. Yardley, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, Nashville, Tennessee, United States

REFERENCES:
- [Result] Yardley DA, Burris HA 3rd, Simons L, Spigel DR, Greco FA, Barton JH, Shipley D, Drosick D, Hainsworth JD. A phase II trial of gemcitabine/carboplatin with or without trastuzumab in the first-line treatment of patients with metastatic breast cancer. Clin Breast Cancer. 2008 Oct;8(5):425-31. doi: 10.3816/CBC.2008.n.051. PMID 18952556
- See also: Published article in Clinical Breast Cancer — http://cigjournals.metapress.com/content/g08721000w0x7572/fulltext.pdf